CLINICAL TRIAL: NCT03074097
Title: Effect of Rectus Sheath Block on Opioid Consumption and Serum Level of TNF-α and IL-6 After Radical Prostatectomy
Brief Title: Rectus Sheath Block: Postoperative Analgesia and Proinflammatory Cytokines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrady S Ibrahim, MD, Assistant professor of anesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 17100391
Record Dates: First submitted 2017-02-27; First posted 2017-03-08 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Postoperative Pain
Keywords: Rectus sheath block, Postoperative pain,TNF alpha and IL-6
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rectus Sheath (Active Comparator): Each patient received bilateral single shot ultrasound guided rectus sheath block under complete aseptic condition in a dose of 30 ml of bupivacaine 0.25% in each side immediately after induction of general anaesthesia
  Interventions: Drug: Bupivacaine 0.25%
- Control (No Intervention): Control group: the patients did not receive any intervention after anaesthesia induction.

INTERVENTIONS:
Drug: Bupivacaine 0.25% — Each patient received bilateral single shot ultrasound guided rectus sheath block under complete aseptic condition in a dose of 30 ml of bupivacaine 0.25% in each side immediately after induction of general anaesthesia
  Other Names: Plain marcaine
  Arms: Rectus Sheath

SUMMARY:
Good quality of postoperative analgesia would lead to attenuate or prevent the adverse effects on the common functions of the immune system. We compared the effect of epidural analgesia versus rectus sheath block on postoperative pain and proinflammatory cytokines following malignant urological surgery.

DETAILED DESCRIPTION:
Study groups: 60 patients were included in the study randomly allocated into two groups of 30 patients. Rectus sheath group (RSB): Each patient received bilateral single shot ultrasound guided rectus sheath block under complete aseptic condition in a dose of 30 ml of bupivacaine 0.25% in each side immediately after induction of general anaesthesia. Control group: the patients did not receive any intervention after anaesthesia induction.

ELIGIBILITY:
Inclusion Criteria:

Male patients their age over 40 years, classified ASA I, II or III, undergoing radical resection of cancer prostate, through midline abdominal incision under general anaesthesia.

Exclusion criteria:

Contraindications to rectus sheath block as patient refusal, coagulopathy, local infection and allergy to bupivacaine. Planned transverse or oblique abdominal incision, extensive existing midline abdominal scarring or pre-existing chronic abdominal pain.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03-05 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2016-04-28 (Actual)

PRIMARY OUTCOMES:
cumulative opioid consumption | 24 hours postoperative
  study the effect of RSB on cumulative opioid consumption at 24 hours

SECONDARY OUTCOMES:
Numerical rating scale (NRS) | 24 hours postoperative
  evaluate postoperative pain intensity by NRS
time to first anlgesic request | 24 hours postoperative
  the first time receiving IV-PCA bolus injection
serum levels of TNF-α | at 24 hours postoperative
  Proinflamatory cytokines
Serum level of IL-6 | at 24 hours postoperative
  Proinflamatory cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Waleed S Farrag, Principal Investigator — Assiut University
Locations (1):
- Assiut university faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hong JY, Lim KT. Effect of preemptive epidural analgesia on cytokine response and postoperative pain in laparoscopic radical hysterectomy for cervical cancer. Reg Anesth Pain Med. 2008 Jan-Feb;33(1):44-51. doi: 10.1016/j.rapm.2007.07.010. PMID 18155056